CLINICAL TRIAL: NCT02478970
Title: Comparison of Clinical Evaluation of Endothelial Cells With Paracentral and Central Specular Microscopy
Brief Title: Specular Microscopy Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment/software did not work as anticipated
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shahzad Mian, Terry J Bergstrom Collegiate Professor of Resident Education in Ophthalmology and Visual Sciences and Associate Professor of Oph, Ophthalmology & Visual Science, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00087911
Record Dates: First submitted 2015-04-24; First posted 2015-06-23 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Endotheliopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corneal endotheliopathy (Experimental): Patients with primary corneal endotheliopathies, such as posterior polymorphous dystrophy, congenital hereditary endothelial dystrophy, Fuchs' dystrophy, iridocorneal endothelial syndrome will be evaluated with the NIDEK CEM-350 and Konan SP4000
  Interventions: Device: Konan SP4000; Device: NIDEK CEM-350
- Normal (Placebo Comparator): Patients without corneal endotheliopathies will be evaluated with the NIDEK CEM-350 and Konan SP4000
  Interventions: Device: Konan SP4000; Device: NIDEK CEM-350

INTERVENTIONS:
Device: Konan SP4000 — current standard of care at Kellogg Eye Center
Device: NIDEK CEM-350 — newly marketed device

SUMMARY:
The corneal endothelium plays an important role in regulating stromal hydration and maintaining the transparency of the cornea. For evaluating the cornea, the most important parameters are corneal endothelial morphology and central corneal thickness. The specular microscope does this. The image in specular microscope is obtained by the specular reflex at a regular, smooth-surfaced interface of two refractive indices, with the angle of the light passing into the cornea equal to the angle of reflection to the observer. To obtain a clear image, the endothelial apical surface must be smooth and uniform and the cornea must be transparent. Nowadays different types of specular microscope exist.

The investigators propose to compare the endothelial cells with two specular microscopes: the Konan SP4000, which is the current model and used for standard of care, to the Nidek CEM-350, which is a newly marketed device.

The investigators would like to evaluate the patients in the clinic and have assessments completed with both specular microscopes.

Nidek will be loaning the specular microscope, NIDEK CEM-530, for the study.

DETAILED DESCRIPTION:
Subjects that provide informed consent will be clinically evaluated (visual acuity, refraction, slit-lamp biomicroscopy, tonometry) by a corneal specialist. After endothelium evaluation with use of slit-lamp biomicroscopy a grade of severity will be given. The grades will be based on the density and confluence of guttae and presence of clinical edema.

Two microscopes, non-contact specular microscope (KONAN SP4000) and paracentral non-contact specular microscope (NIDEK CEM-350), will be used for the exam.

For each patient both eyes will be examined by the two non-contact specular microscopes.

Three pictures of the central cornea will be captured from the standard specular microscope.

The paracentral specular microscope can capture image of one central point, eight paracentral points with 5° visual angle and six peripheral points with 27° visual angle. It will capture 16 images and automatically will classify based on quality and the ability to be analyzed. The optimal image for analysis will be indicated with orange highlight. Once the image is selected, a new manual or automatic software will be used to count the endothelial cells, complete analysis will be automatically performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older;
* Patients with primary corneal endotheliopathies (posterior polymorphous dystrophy, congenital hereditary endothelial dystrophy, Fuchs' dystrophy, iridocorneal endothelial syndrome;
* Healthy patients without corneal endotheliopathies.

Exclusion Criteria:

* Patients with history of corneal and/or intraocular surgery;
* Patients with existing corneal and/or anterior segment disease, except for the inclusion criteria;
* Intraocular pressure ≥21mmHg;
* Contact lens wearer;
* History of ocular trauma;
* Patients with diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Endothelial cell count | Approximately at the end of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Mian, MD, Principal Investigator — University of Michigan Kellogg Eye Center
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No